CLINICAL TRIAL: NCT00704002
Title: Conservative Versus Operative Treatment of Displaced Neck Fractures of the Fifth Metacarpal
Acronym: CONFraM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONFraM
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Fifth Metacarpal Neck Fracture
Keywords: neck fracture of the fifth metacarpal; displacement; antegrade intramedullary splinting; conservative treatment
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): antegrade intramedullary splinting
  Interventions: Procedure: antegrade intramedullary splinting
- B (Active Comparator): conservative treatment
  Interventions: Procedure: conservative treatment

INTERVENTIONS:
Procedure: antegrade intramedullary splinting — antegrade intramedullary splinting with 2 to 3 small K-wires
  Arms: A
Procedure: conservative treatment — conservative treatment with 2-finger splint for one week
  Arms: B

SUMMARY:
This is a prospective, randomized, multi-center pilot study of isolated, displaced neck fractures of the fifth metacarpal. The patients are randomly assigned to osteosynthesis with antegrade intramedullary splinting or conservative treatment.

DETAILED DESCRIPTION:
The aim of this study is to provide criteria for treatment decisions in patients with isolated, displaced neck fractures of the fifth metacarpal. The primary outcome criterion is the functional status measured by the Disability of the Arm, Shoulder and Hand (DASH) questionnaire. Secondary outcome criteria are pain, range of motion (ROM), grip strength, and radiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* displaced neck fracture of the fifth metacarpal (at least 30° angulation)
* isolated injury
* age between 18 and 75 years
* informed consent

Exclusion Criteria:

* rotational displacement
* open fracture
* injury older than one week
* treatment other than within this study
* other relevant injuries of the upper extremities
* other injury or disease of the hand
* pregnancy
* missing informed consent
* incompliance
* coagulopathy
* allergy to metallic implants
* Patients who have participated in any other device or drug clinical trial within the previous month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-12; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Disability of the Arm, Shoulder and Hand (DASH) questionnaire | 3 months

SECONDARY OUTCOMES:
pain | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schädel-Höpfner, MD, Principal Investigator — Department of Trauma and Hand Surgery, University Hospital, Düsseldorf, Germany
Locations (1):
- Department of Trauma and Hand Surgery, Düsseldorf, Germany